CLINICAL TRIAL: NCT05140590
Title: Pharmacological Interactions Between Antihypertensive Regimens and Drugs Prescribed in the Emergency Department of the HGZ 51
Brief Title: Interactions Between Antihypertensive Drugs and Drugs Prescribed in the Emergency Room
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Lilia Edith Luque Esparza, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: R-2020-902-030
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Drug Interactions; Hypertension
Keywords: Hypertension; Drug Interactions; Drugs in the emergency room; Antihypertensive Agents
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with a diagnosis of hypertension admitted to the emergency department: Direct questioning about general data, medical history and about the pharmacological scheme for the treatment of hypertension.
  Review of clinical records to obtain data about the admission diagnosis, drugs administered during their hospital stay, and blood pressure figures at admission, during hospital stay and at discharge.
  Analysis and classification of theoretical drug interactions using the IBM Micromedex Drug Interactions and iDoctus clinical decision support systems.

SUMMARY:
Drug interactions (IFF) are events that occur when multiple drugs are administered at the same time to an individual. People with arterial hypertension generally require therapeutic regimens based on 2 or more drugs for their adequate control, which makes them patients with polypharmacy. When these patients require urgent medical attention, there is a risk that IFFs will occur between their base treatment and the drugs that are prescribed to solve the added condition.

Objective. To determine the frequency of pharmacological interactions between antihypertensive regimens and drugs used in the emergency service of Hospital General de Zona No 51 (HGZ 51).

Material and methods: Observational, descriptive, and prospective study. The participants will be eligible patients with systemic arterial hypertension treated in the emergency room of HGZ 51 in Gómez Palacio, Durango. Support systems will be used for clinical decision, to identify potential IFFs and to be able to classify them according to their mechanism (pharmacokinetics and pharmacodynamics) and severity. A descriptive statistical analysis will be carried out in the SPSS program using measures of frequency, dispersion and central tendency.

DETAILED DESCRIPTION:
The researchers will invite individuals with high blood pressure who come to the emergency department in the period from January 2021 to December 2021 to participate in the study. They will be questioned about the selection criteria, and if they are eligible to be included in the study, they will be provided with the informed consent letter for reading, clarification of doubts and signature. Each participant will receive a copy of the informed consent letter.

Participants will be questioned directly to obtain information about their general data, medical history and about their drug treatment for hypertension. The rest of the data (admission diagnosis, drugs administered during their hospital stay, etc.) will be obtained from the clinical record, as well as the blood pressure measurements on admission, during their hospital stay and upon discharge. The analysis of the theoretical pharmacological interactions and their classification will be carried out prior to feeding the database using the IBM Micromedex Drug Interactions and iDoctus Clinical Decision Support Systems (CDSS).

The information obtained will be emptied into an Excel database for subsequent statistical analysis with the SPSS 21 program. The study information will remain confidential under the responsibility of the responsible researcher. As a protection measure on the information collected for the investigation, the personal identification data will be substituted by folio numbers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of arterial hypertension confirmed that they are hospitalized in the emergency department of HGZ 51.
* Pharmacological treatment already established to control hypertension.
* Accept to participate and sign the informed consent.
* Prescription and / or administration of additional drugs to your antihypertensive treatment during your hospital stay in the emergency department.

Exclusion Criteria:

* That they do not know or do not provide complete information on their basic antihypertensive treatment.

Elimination criteria

* Survey with incomplete pharmacotherapeutic history data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Beneficiaries with a history of a diagnosis of arterial hypertension who are hospitalized in the emergency service of the HGZ 51.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of theoretical IFFs detected | Duration of hospitalization (15 days)
  Potential for the prescription of a drug associated with other active ingredients to generate a risk of drug interaction.
  Number of theoretical IFFs detected by support systems for clinical decision
Frequency of IFF by pharmacological mechanism | Duration of hospitalization (15 days)
  Number of interactions detected by support systems for clinical decision classified according to the pharmacological mechanism into pharmacokinetics or pharmacodynamics.
  The interactions of absorption, distribution, metabolism and excretion will be considered pharmacokinetic.
  Interactions by synergy (addition, potentiation), antagonism, hypersensitization and desensitization will be considered pharmacodynamic.
Degree severity of drug interaction detected | Duration of hospitalization (15 days)
  Classification of IFFs according to the theoretical severity provided by the support systems for clinical decision.
  1. Minors (without clinical condition)
  2. Moderate (may cause deterioration of clinical status)
  3. Major (can be life-threatening or cause permanent damage)
  4. Contraindicated (should not be used simultaneously)

SECONDARY OUTCOMES:
Control of hypertension according to blood pressure figures at admission | upon admission (2 horas)
  According to the provisions of the 2018 ESC/ESH Guide on the diagnosis and treatment of arterial hypertension, blood pressure figures are considered to be control at admission to the emergency room of:
  Systolic blood pressure (SBP) <140 mmHg Diastolic blood pressure (DBP) <90 mmHg
Control of hypertension according to blood pressure figures during hospitalization | Duration of hospitalization (15 days)
  According to the provisions of the 2018 ESC/ESH Guide on the diagnosis and treatment of arterial hypertension, blood pressure figures are considered to be control during hospitalization to the emergency room of:
  SBP <140 mmHg DBP <90 mmHg
Control of hypertension according to blood pressure figures at discharge | At the time of discharge (2-15 days)
  In accordance with the provisions of the 2018 ESC/ESH Guide on the diagnosis and treatment of arterial hypertension, blood pressure figures are considered controlled upon discharge from hospitalization in the emergency department of:
  SBP <140 mmHg DBP <90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Lilia E Luque-Esparza, Dra., Principal Investigator — IMSS
Locations (1):
- Instituto Méxicano del Seguro Social HGZ No.51, Gómez Palacio, Durango, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
This item has not yet been defined

REFERENCES:
- [Background] Amariles P, Giraldo NA, Faus MJ. [Clinical relevance of drug interactions]. Med Clin (Barc). 2007 Jun 2;129(1):27-35. doi: 10.1157/13106681. Spanish. PMID 17570184
- [Background] Iniesta-Navalon C, Urbieta-Sanz E, Gascon-Canovas JJ. [Analysis of the drug interactions associated to domiciliary drug therapy in elderly hospitalized patients]. Rev Clin Esp. 2011 Jul-Aug;211(7):344-51. doi: 10.1016/j.rce.2011.04.005. Epub 2011 Jun 2. Spanish. PMID 21640341
- [Background] Horn JR, Hansten PD, Chan LN. Proposal for a new tool to evaluate drug interaction cases. Ann Pharmacother. 2007 Apr;41(4):674-80. doi: 10.1345/aph.1H423. Epub 2007 Mar 27. PMID 17389673
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Morales-Olivas FJ, Estan L. [Antihypertensive drug-drug interactions]. Med Clin (Barc). 2005 May 28;124(20):782-9. doi: 10.1157/13075851. Spanish. PMID 15927106
- See also: Guía de práctica clínica de interacciones farmacológicas potenciales en la atención del adulto mayor — http://www.imss.gob.mx/sites/all/statics/guiasclinicas/688GER.pdf
- See also: Drug Interactions in hospitalized patients in the Internal Medicine Hospital University " Dr. Angel Larralde ". June 2014 - December 2015 — http://ve.scielo.org/scielo.php?script=sci_arttext&pid=S0798-02642016000100001&lng=es.
- See also: Guía de Práctica Clínica Prescripción farmacológica razonada para el adulto mayor — http://www.imss.gob.mx/sites/all/statics/guiasclinicas/558GER.pdf